CLINICAL TRIAL: NCT05527756
Title: Evaluation of the Cosmetic Outcomes of Totally Endoscopic Cardiac Surgery
Acronym: SCARMICS
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: f/2022/121
Record Dates: First submitted 2022-08-31; First posted 2022-09-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Minimally Invasive Cardiac Surgery; Scar
MeSH Terms: conditions — Cicatrix | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Totally endoscopic aortic/mitral valve replacement: Study procedures include the Scar Cosmesis Assessment and Rating (SCAR) scale and numerical rating scale (NRS) questionnaire at one, 14 and 30 days after totally endoscopic aortic/mitral valve replacement. Additionally, a photo of the incisions will be taken at these time points.
  Interventions: Other: Scar Cosmesis Assessment and Rating (SCAR) scale; Other: Numerical rating scale (NRS)
- Totally endoscopic coronary artery bypass grafting: Study procedures include the Scar Cosmesis Assessment and Rating (SCAR) scale and numerical rating scale (NRS) questionnaire at one, 14 and 30 days after totally endoscopic coronary artery bypass grafting. Additionally, a photo of the incisions will be taken at these time points.
  Interventions: Other: Scar Cosmesis Assessment and Rating (SCAR) scale; Other: Numerical rating scale (NRS)

INTERVENTIONS:
Other: Scar Cosmesis Assessment and Rating (SCAR) scale — The SCAR scale consists of two simple questions about symptoms (itch and pain) with yes/no response options that are responded to by the patient and six clinician-related items that are rated by observers through photos of the incisions. This scale includes both objective measurements and patient-reported symptoms
Other: Numerical rating scale (NRS) — The NRS scale, in which the patients score the cosmetic appearance of the scar from 0 to 10, is questioned.

SUMMARY:
Totally endoscopic cardiac surgery (TECS) is considered to have aesthetic advantages over conventional median sternotomy due to the smaller incisions. Most research regarding TECS focuses on clinical outcomes instead of cosmetic consequences. Following surgery, postoperative scarring is unavoidable and may negatively affect the patient's physical and emotional well-being. Therefore, this study aims to investigate the cosmesis after TECS.

DETAILED DESCRIPTION:
Totally endoscopic cardiac surgery (TECS) is considered to have aesthetic advantages over conventional median sternotomy due to the smaller incisions. Most research regarding TECS focuses on clinical outcomes instead of cosmetic consequences. Following surgery, postoperative scarring is unavoidable and may negatively affect the patient's physical and emotional well-being. One previous study compared median sternotomy cardiac surgery and TECS in terms of the long-term cosmetic appearance of postoperative scars. They concluded that scars were considered more satisfactory, less painful, and itchy in the TECS group in the Chinese population. To our knowledge, this is the only study published regarding cosmetic consequences after TECS. Therefore, this study aims to investigate the cosmesis after TECS.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Patients who can give their informed consent
* Patients who speak Dutch or French

Exclusion Criteria:

* Patients that previously underwent cardiac surgery
* Patients that will undergo a combination of cardiac surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that undergo totally endoscopic aortic valve replacement (TEAVR), totally endoscopic mitral valve (MVATS) and totally endoscopic coronary artery bypass grafting (Endo-CABG) at the Department of Cardiothoracic Surgery of the Jessa Hospital, Hasselt will be screened for eligibility.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2023-05-27 (Actual); Study Completion 2023-05-27 (Actual)

PRIMARY OUTCOMES:
Evaluate the cosmesis through the Scar Cosmesis Assessment and Rating (SCAR) scale at postoperative day one. | Postoperative day one
  The SCAR scale includes both objective measurements and patient-reported symptoms. A low score corresponds to a good scar cosmesis and a high score to a bad scar cosmesis.
Evaluate the cosmesis through the Scar Cosmesis Assessment and Rating (SCAR) scale at postoperative day 14. | Postoperative day 14
  The SCAR scale includes both objective measurements and patient-reported symptoms. A low score corresponds to a good scar cosmesis and a high score to a bad scar cosmesis.
Evaluate the cosmesis through the Scar Cosmesis Assessment and Rating (SCAR) scale at postoperative day 30. | Postoperative day 30
  The SCAR scale includes both objective measurements and patient-reported symptoms. A low score corresponds to a good scar cosmesis and a high score to a bad scar cosmesis.

SECONDARY OUTCOMES:
Cosmetic assessment from the patients through the numerical rating scale (NRS) at postoperative day one. | Postoperative day one
  The cosmetic appearance of the scar is scored from 0 to 10, whereas 0 contributes to not satisfied with the scar and 10 with very satisfied with the scar.
Cosmetic assessment from the patients through the numerical rating scale (NRS) at postoperative day 14. | Postoperative day 14
  The cosmetic appearance of the scar is scored from 0 to 10, whereas 0 contributes to not satisfied with the scar and 10 with very satisfied with the scar.
Cosmetic assessment from the patients through the numerical rating scale (NRS) at postoperative day 30. | Postoperative day 30
  The cosmetic appearance of the scar is scored from 0 to 10, whereas 0 contributes to not satisfied with the scar and 10 with very satisfied with the scar.

CONTACTS AND LOCATIONS:
Overall Officials: Alaaddin Yilmaz, MD, Study Chair — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No